CLINICAL TRIAL: NCT00579527
Title: Phase I/II Trial of Thymus Transplantation With Immunosuppression, #950
Brief Title: Phase I/II Thymus Transplantation With Immunosuppression #950
Acronym: #950
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011583; 2R01AI047040-11A2 (NIH); R56 Bridge R01AI4704011A1 (Other Grant/Funding Number: [NIH American Recovery and Reinvestment Act (ARRA) of 2009]); 5K12HD043494-09 (NIH); R01AI047040 (NIH); R01AI054843 (NIH); 950 (Other: Duke)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: DiGeorge Anomaly; Complete DiGeorge Anomaly; Complete Atypical DiGeorge Anomaly; Complete DiGeorge Syndrome; Complete Atypical DiGeorge Syndrome
Keywords: DiGeorge Anomaly; Thymus Transplantation; DiGeorge Syndrome; Athymia; Parathyroid Transplantation; Hypocalcemia; Hypoparathyroidism; Low T cell numbers; Immunoreconstitution; Immunodeficiency; Complete DiGeorge Anomaly; Complete Atypical DiGeorge Anomaly; Complete DiGeorge Syndrome; Complete Atypical DiGeorge Syndrome; Cultured Thymus Tissue Implantation (CTTI)
MeSH Terms: conditions — DiGeorge Syndrome; Thymic aplasia; Hypocalcemia; Hypoparathyroidism; Immunologic Deficiency Syndromes | interventions — Drug Implants; Thymus Extracts; Blood Specimen Collection; Phlebotomy; Antilymphocyte Serum; thymoglobulin; Cyclosporine; Cyclosporins; Tacrolimus; Methylprednisolone; Prednisolone; Steroids; Daclizumab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cultured Thymus Tissue Implantation (CTTI) w/immunosuppression (Experimental): Patients with complete DiGeorge Anomaly (cDGA) undergo cultured thymus tissue implantation (previously described as transplantation) with tailored immunosuppression based on the subject's pre-implantation T cell numbers and function.
  Interventions: Biological: Cultured Thymus Tissue for Implantation (CTTI); Procedure: Blood Draw; Drug: Rabbit anti-thymocyte globulin; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Methylprednisolone or Prednisolone; Drug: Daclizumab; Drug: Mycophenolate mofetil
- CTTI with Parathyroid Transplantation w/immunosuppression (Experimental): Patients with complete DiGeorge Anomaly (cDGA) undergoes cultured thymus tissue thymus implantation (previously described as transplantation) with tailored immunosuppression based on the subject's pre-implantation T cell numbers and function. If the patient has hypoparathyroidism, and is eligible, the patient may also receive a parathyroid transplant.
  Interventions: Other: Cultured Thymus Tissue Implantation and Parental Parathyroid Transplantation; Procedure: Blood Draw; Drug: Rabbit anti-thymocyte globulin; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Methylprednisolone or Prednisolone

INTERVENTIONS:
Biological: Cultured Thymus Tissue for Implantation (CTTI) — Potential thymus recipient subjects are screened for eligibility. Thymus donor (unrelated donor), and thymus donor's birth mother are screened for safety. CTTI is done under general anesthesia in the operating room. Cultured thymus tissue is implanted into the subject's quadriceps. Two to three months post CTTI, if medically stable, the subject undergoes allograft biopsy. At the time of implantation and biopsy, a skin biopsy is done. Immunosuppression is weaned as per protocol.
  Other Names: Thymus Tissue Transplant; CTTI
  Arms: Cultured Thymus Tissue Implantation (CTTI) w/immunosuppression
Other: Cultured Thymus Tissue Implantation and Parental Parathyroid Transplantation — For subjects w/ hypoparathyroidism, the subject may receive CTTI and parathyroid transplant. For parathyroid transplant, parental parathyroid donors are screened. Parathyroid is harvested from the parent who shares the most Human Leukocyte Antigens (HLA) alleles with the thymus donor. Parathyroid gland is minced and placed in quadriceps muscle; there is no dose. Parathyroid donors are monitored as outpatients until recipients' discharge. Recipients' calcium and PTH levels are monitored indefinitely. Potential thymus recipient subjects are screened for eligibility. Thymus donor (unrelated donor), and thymus donor's birth mother are screened for safety. CTTI is done under general anesthesia in the operating room. Cultured thymus tissue is implanted into the subject's quadriceps. Two to three months post CTTI, if medically stable, the subject undergoes allograft biopsy. At the time of CTTI and biopsy, a skin biopsy is done. Immunosuppression is weaned as per protocol.
  Other Names: Thymus and Parathyroid Transplant; CTTI and Parathyroid Transplant
  Arms: CTTI with Parathyroid Transplantation w/immunosuppression
Procedure: Blood Draw — Birth mothers of Thymus Recipients are asked to participate in the study and undergo phlebotomy to allow testing of T cell identity in the Complete DiGeorge subjects. If blood is not obtainable then a buccal swab may be done.
  Other Names: Venipuncture
Drug: Rabbit anti-thymocyte globulin — Three doses of 2 mg/kg IV (through a central venous catheter) prior to CTTI. Each dose of Rabbit anti-thymocyte globulin (RATGAM) is given over 12 hours. RATGAM is usually given on days-5, -4, and -3 prior to CTTI or CTTI and parathyroid transplantation. Medications (diphenhydramine, steroids, and acetaminophen) are given with rabbit anti-thymocyte globulin.
  Other Names: RATGAM; thymoglobulin
Drug: Cyclosporine — In addition to RATGAM, subjects with typical cDGA with PHA responses >50,000 cpm, or atypical cDGA with PHA response <75,000cpm (when not on immunosuppression) or <40,000 cpm to PHA while on immunosuppression, are started on cyclosporine (Csa) as soon as cDGA is diagnosed. Csa is continued with target trough levels of 180 to 220 ng/ml. If subject cannot tolerate Csa, Csa may be changed to tacrolimus (FK506) with target trough level 7 to 10 ng/ml. When trough levels are outside of range, dosing is modified appropriately.
  Csa may be given every 8 to 12 hours enterally or IV before and after CTTI. The Csa dose is dependent on T cell numbers and the target Csa trough levels. Csa is weaned as per protocol.
  Other Names: Csa
Drug: Tacrolimus — If unable to tolerate cyclosporine, then tacrolimus is given. Tacrolimus may be given every 8 to 12 hours enterally or IV before and after the CTTI transplant. Tacrolimus dose is dependent on the T cell numbers and the target tacrolimus trough levels. Tacrolimus is weaned as per protocol.
  Other Names: FK506
Drug: Methylprednisolone or Prednisolone — Steroids IV or enterally may be given before and after CTTI or CTTI and parathyroid transplantation. Administration and dosage depends on T cell numbers and symptoms. Pre-transplant steroids may be used when pre-transplant T cells >4,000cumm. Steroids are weaned as per protocol.
  Other Names: Steroids
Drug: Daclizumab — In addition, subjects with Atypical DiGeorge with PHA responses >75,000cpm while on no immunosuppression or PHA responses >40,000cpm while on immunosuppression, Daclizumab 1 mg/kg single dose IV may be given depending on T cell counts. Administration of Daclizumab depends on T cell numbers and T cell activation. A single dose may be given after the administration of rabbit anti-thymocyte globulin and before CTTI. If Daclizumab is not given before CTTI, and, depending on the T cell numbers and T cell activation, a single dose of Daclizumab may be given 3-5 days after CTTI.
  Other Names: Zenapax
  Arms: Cultured Thymus Tissue Implantation (CTTI) w/immunosuppression
Drug: Mycophenolate mofetil — In addition, subjects with Atypical DiGeorge with PHA responses >75,000cpm while on no immunosuppression or PHA responses >40,000cpm while on immunosuppression, Mycophenolate mofetil 15 mg/kg/dose every 8 hours IV or enterally may be given depending on T cell counts. Mycophenolate mofetil may be given if the T cell count remains elevated 5 days after CTTI. If MMF is given, the dose is 15 mg/kg IV. MMF may be stopped at 35 days after CTTI or continued for up to six months after CTTI.
  Other Names: MMF; CellCept
  Arms: Cultured Thymus Tissue Implantation (CTTI) w/immunosuppression

SUMMARY:
The study purpose is to determine if cultured thymus tissue implantation (CTTI) (previously described as transplantation) with tailored immunosuppression based on the recipient's pre-implantation T cell population is a safe and effective treatment for complete DiGeorge anomaly. This study will also evaluate whether cultured thymus tissue implantation and parathyroid transplantation with immunosuppression is a safe and effective treatment for complete DiGeorge anomaly and hypoparathyroidism.

DETAILED DESCRIPTION:
Complete DiGeorge anomaly is a congenital disorder characterized by athymia. Without successful treatment, children remain immunodeficient and usually die by age 2 years. In infants with complete DiGeorge anomaly and no T cells, cultured thymus tissue implantation (CTTI) without immunosuppression resulted in diverse T cell development and good T cell function. Some infants with no thymus have some T cells that presumably developed extrathymically; these T cells can reject a thymus graft.

The purpose of this study is to tailor immunosuppression use for complete DiGeorge anomaly subjects who have some T cells and different T cell function levels. This protocol includes tailored immunosuppression regimens to allow subjects with different T cell function levels to be suppressed adequately.

Patients with complete DiGeorge often have hypoparathyroidism, a life threatening condition. Successful CTTI does not result in improvement of the hypoparathyroidism. The patients must go to the clinic for frequent calcium levels and to the hospital for calcium infusions. These infants are at risk for seizures from low calcium. This study had a parental parathyroid transplant arm for subjects with hypoparathyroidism who require calcium replacement.

Whether or not a subject was enrolled in the parathyroid arm, the immunosuppression regimen the subject received was dependent on the immune findings as stated in the clinical protocol.

ELIGIBILITY:
Thymus Transplantation Inclusion:

* Must have 1 of following: 22q11 or 10p13 hemizygosity; hypocalcemia requiring replacement; congenital heart defect; CHARGE association or CHD7 mutation; or abnormal ears plus mother w/diabetes (type I, type II, gestational).
* <50 CD3+ T cells/cumm or <50 CD3+ T cells/cumm that are CD62L+ CD45RA+ (cluster of differentiation 45RA) (naïve phenotype), or <5% of CD3+ count being CD62L+ CD45RA+

Atypical DiGeorge:

* Must have, or have had, a rash. If rash present, rash biopsy must show T cells in skin. If rash & adenopathy resolved, must have >50/cumm T cells & naive T cell must be <50/cumm or <5% of T cells.

Typical DiGeorge:

* CD3+ CD45RA+ CD62L+ T cells <50/mm3 or <5% of total T cells

Parathyroid Transplantation Additional Inclusion:

* 2 studies in recipient which PTH<5 pg/ml when ionized calcium <1.1 mmol/L. Can be done anytime pre-tx; 1 must be done while at Duke Hospital.
* Parent(s) willing & eligible to be donors

Thymus Transplantation Exclusion:

* Heart surgery <4 wks pre-tx
* Heart surgery anticipated w/in 3 months after proposed tx
* Rejection by surgeon or anesthesiologist as surgical candidate
* Lack of sufficient muscle tissue to accept transplant of 4 grams/m2 BSA
* HIV infection
* Prior attempts at immune reconstitution, such as bone marrow tx or previous thymus tx
* CMV(>500 copies/ml blood by PCR on 2 tests)
* Ventilator dependence

Parathyroid Donor Inclusion:

* >18 years of age
* Serum calcium in normal range
* Normal PTH function
* HLA typing consistent with parentage
* Not on anticoagulation or can come off
* Parent chosen will share HLA-DR allele with thymus donor that was not inherited by the recipient. If no HLA matching at all, then either parent is acceptable if the parent meets other criteria.

Parathyroid Donor Exclusion:

* <18 years old
* Hypoparathyroidism-low PTH in presence of low serum calcium & high serum phosphate
* Hyperparathyroidism(or history)-elevated PTH in presence of high serum calcium and low serum phosphate.
* History of cancer
* Donor only living involved parent/guardian of recipient
* Evidence of HIV-1, HIV-2, HTLV-1, HTLV-2, syphilis, hepatitis B, hepatitis C, West Nile virus, or Chagas disease
* Creutzfeldt Jakob disease (CJD)
* Elevated liver function studies: AST, ALT, alkaline phosphatase >3x upper normal limit
* Receipt of xenograft or risk factors for SARS, CJD and/or smallpox exposure. {If CJD risk factors but not active disease, parent may give permission for parathyroid use.}
* Urine CMV positive
* Positive CMV IgM
* Positive IgM anti-EBV VCA
* On blood thinners and cannot stop for parathyroid donation
* Elevated PT or PTT (>ULN)
* Platelets<100,000
* Positive Toxoplasma IgM
* Donor will receive a history and physical; may be excluded based on PI's medical judgment.
* Hemoglobin <9g/dl
* Infectious head or neck lesion
* Goiter on ultrasound
* Abnormal fiberoptic laryngoscopy of vocal cords
* HLA inconsistent with parentage
* Pregnancy
* Positive HSV IgG isn't exclusion; post-tx prophylaxis needed for recipient if donor is HSV IgG+.
* Positive VZV IgG isn't exclusion; post-tx prophylaxis needed if donor is VZV IgG+.
* Medical concern of independent otolaryngologist.
* Concern by medical psychologist/social worker that potential donor isn't competent or does not understand risks.
* Questionnaire responses can lead to exclusion.

Mother of DiGeorge Inclusion:

• Provides consent to use blood/buccal sample. No exclusions except unwillingness to consent; or, provide blood/buccal sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-12-19 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Louise Markert, MD, PhD, Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Background] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sedlak DA, Sempowski GD, Hale LP, Rice HE, Mahaffey SM, Skinner MA. Postnatal thymus transplantation with immunosuppression as treatment for DiGeorge syndrome. Blood. 2004 Oct 15;104(8):2574-81. doi: 10.1182/blood-2003-08-2984. Epub 2004 Apr 20. PMID 15100156
- [Background] Markert ML and Devlin BH. Thymic reconstitution (in Rich RR, Shearer WT, Fleischer T, Schroeder HW, Weyand CM, Frew A, eds., Clinical Immunology 3rd edn., Elsevier, Edinburgh) p 1253-1262, 2008.
- [Background] Selim MA, Markert ML, Burchette JL, Herman CM, Turner JW. The cutaneous manifestations of atypical complete DiGeorge syndrome: a histopathologic and immunohistochemical study. J Cutan Pathol. 2008 Apr;35(4):380-5. doi: 10.1111/j.1600-0560.2007.00816.x. PMID 18333898
- [Background] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Background] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sempowski GD, Rhein ME, Szabolcs P, Hale LP, Buckley RH, Coyne KE, Rice HE, Mahaffey SM, Skinner MA. Complete DiGeorge syndrome: development of rash, lymphadenopathy, and oligoclonal T cells in 5 cases. J Allergy Clin Immunol. 2004 Apr;113(4):734-41. doi: 10.1016/j.jaci.2004.01.766. PMID 15100681
- [Background] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Background] Li B, Li J, Devlin BH, Markert ML. Thymic microenvironment reconstitution after postnatal human thymus transplantation. Clin Immunol. 2011 Sep;140(3):244-59. doi: 10.1016/j.clim.2011.04.004. Epub 2011 Apr 16. PMID 21565561
- [Background] Chinn IK, Olson JA, Skinner MA, McCarthy EA, Gupton SE, Chen DF, Bonilla FA, Roberts RL, Kanariou MG, Devlin BH, Markert ML. Mechanisms of tolerance to parental parathyroid tissue when combined with human allogeneic thymus transplantation. J Allergy Clin Immunol. 2010 Oct;126(4):814-820.e8. doi: 10.1016/j.jaci.2010.07.016. Epub 2010 Sep 15. PMID 20832849
- [Result] Markert ML, Devlin BH, McCarthy EA. Thymus transplantation. Clin Immunol. 2010 May;135(2):236-46. doi: 10.1016/j.clim.2010.02.007. Epub 2010 Mar 16. PMID 20236866
- [Result] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759
- [Result] Hudson LL, Louise Markert M, Devlin BH, Haynes BF, Sempowski GD. Human T cell reconstitution in DiGeorge syndrome and HIV-1 infection. Semin Immunol. 2007 Oct;19(5):297-309. doi: 10.1016/j.smim.2007.10.002. Epub 2007 Nov 26. PMID 18035553
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA, Li YJ. Factors affecting success of thymus transplantation for complete DiGeorge anomaly. Am J Transplant. 2008 Aug;8(8):1729-36. doi: 10.1111/j.1600-6143.2008.02301.x. Epub 2008 Jun 28. PMID 18557726
- [Result] Markert ML, Devlin BH, McCarthy EA, Chinn IK, Hale LP. Thymus Transplantation in Thymus Gland Pathology: Clinical, Diagnostic, and Therapeutic Features. Eds Lavinin C, Moran CA, Morandi U, Schoenhuber R. Springer-Verlag Italia, Milan, 2008, pp 255-267.
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA. Thymus transplantation in complete DiGeorge anomaly. Immunol Res. 2009;44(1-3):61-70. doi: 10.1007/s12026-008-8082-5. PMID 19066739
- [Result] Chinn IK, Milner JD, Scheinberg P, Douek DC, Markert ML. Thymus transplantation restores the repertoires of forkhead box protein 3 (FoxP3)+ and FoxP3- T cells in complete DiGeorge anomaly. Clin Exp Immunol. 2013 Jul;173(1):140-9. doi: 10.1111/cei.12088. PMID 23607606

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The goal of this study is survival of subjects after cultured thymus tissue implantation (CTTI) regardless of the immunosuppressive regimen or of parathyroid co-transplantation.
Groups:
- Cultured Thymus Tissue Implantation w/ Immunosuppression: Participants enrolled in cultured thymus tissue implantation (CTTI) with immunosuppression were given immunosuppression based on results of flow cytometry without consideration of whether a parathyroid transplant would be given.
  No participants were enrolled into Arm 2. No subjects received a parathyroid transplant.
  No specific dose of cultured thymus tissue was assigned. The dose was the number of grams of cultured thymus tissue divided by the weight of the recipient in kg or per square meter of body surface area of the participant.
  There was one administration of cultured thymus tissue. The dosage form was cultured thymus tissue.
Period: Overall Study
Arm/Group | Cultured Thymus Tissue Implantation w/ Immunosuppression
Started | 14
Completed | 10
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Groups:
- Cultured Thymus Tissue Implantation With Immunosuppression: Participants enrolled into cultured thymus tissue for implantation (previously described as transplantation) with immunosuppression were given immunosuppression based on the subject's pre-implantation T cell number and function.
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 248 (161)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8
  Black or African American | 3
  American Indian or Alaska Native | 2
  More than One Race (Caucasian/Asian) | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Survival at 1 Year Post-CTTI
Description: Survival at 1 year post cultured thymus tissue implantation was assessed using the Kaplan Meier Estimated Survival. This mathematical function estimates the survival for a certain length of time.
Time Frame: 1 year post-CTTI
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: % of participants who survive to 1 year
Groups:
- Cultured Thymus Tissue With Immunosuppression: Participants enrolled into cultured thymus tissue for Implantation (previously described as transplantation) with immunosuppression were given immunosuppression based on the subject's pre-implantation T cell numbers and function.
Arm/Group | Cultured Thymus Tissue With Immunosuppression
Number analyzed (Participants) | 14
% of participants who survive to 1 year | 71 [40.6 to 88.2]

2. Secondary Outcome: Survival at 2 Years Post-CTTI
Description: Survival at 2 years post cultured thymus tissue implantation was assessed using the Kaplan Meier Estimated Survival. This mathematical function estimates the survival for a certain length of time.
Time Frame: 2 years post-CTTI
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: % of participants who survive to 2 years
Groups:
- Cultured Thymus Tissue Implantation With Immunosuppression: Participants enrolled into Cultured Thymus Tissue Implantation (previously described as transplantation) with immunosuppression were given immunosuppression based on the subject's pre-implantation T cell numbers and function.
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 14
% of participants who survive to 2 years | 71 [40.6 to 88.2]

3. Secondary Outcome: Immune Reconstitution Efficacy - Total CD3 T Cells
Description: The development of total CD3 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included for the 1 year time point if a CD3 T cell count was performed in relevant time period. The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 9
cells/mm3 | 726 [345 to 1866]

4. Secondary Outcome: Immune Reconstitution Efficacy - Total CD4 T Cells
Description: The development of total CD4 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included for the 1 year time point if a CD4 T cell count was performed in relevant time period. The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 10
cells/mm3 | 593 [230 to 1780]

5. Secondary Outcome: Immune Reconstitution Efficacy - Total CD8 T Cells
Description: The development of total CD8 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included for the 1 year time point if a CD8 T cell count was performed in relevant time period. The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 10
cells/mm3 | 145 [22 to 360]

6. Secondary Outcome: Immune Reconstitution Efficacy - Naive CD4 T Cells
Description: The development of total naive CD4 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included for the 1 year time point if a T cell count was performed in relevant time period. The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 9
cells/mm3 | 156 [23 to 751]

7. Secondary Outcome: Immune Reconstitution Efficacy - Naive CD8 T Cells
Description: The development of total naive CD8 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included for the 1 year time point if a T cell count was performed in the relevant time period. The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 9
cells/mm3 | 37 [4 to 217]

8. Secondary Outcome: Immune Reconstitution Efficacy - Response to Mitogens
Description: Measurement of the T cell proliferative response to the mitogen phytohemagglutin (PHA).
Time Frame: 1 year post-CTTI
Population: Data were only included for the 1 year time point if a testing was performed in the relevant time period. The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Measure: Median (Full Range); unit: counts per minute (cpm)
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 8
counts per minute (cpm) | 139189 [13726 to 202132]

9. Secondary Outcome: Thymus Allograft Biopsy
Description: Evidence, on biopsy of the thymus tissue implanted in muscle, that shows the development of new T cells.
Time Frame: 2 to 3 months post-CTTI
Population: Data were only included if the participant had a biopsy of the thymus tissue implanted. The study was designed to assess survival, without regard to the immune suppression used. No participants were enrolled into Arm 2. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
Number analyzed (Participants) | 10
Participants
  Evidence of thymopoiesis | 7
  Evidence of rejection | 0
  Inconclusive for thymopoiesis | 3

ADVERSE EVENTS:
Time Frame: 2 years post-CTTI
Description: Participants enrolled into Cultured Thymus Tissue for Implantation (previously described as transplantation) with immunosuppression were given immunosuppression based on the subject's pre-implantation T cell numbers and function. All adverse events are reported below.
Groups:
- Cultured Thymus Tissue Implantation With Immunosuppression: Participants enrolled into Cultured Thymus Tissue Implantation (previously described as transplantation) with immunosuppression were given immunosuppression based on the subject's pre-implantation T cell numbers and function. All adverse events were combined for this analysis regardless of the immunosuppression used.
Arm/Group | Cultured Thymus Tissue Implantation With Immunosuppression
All-Cause Mortality (participants affected / at risk) | 4/14
Serious Adverse Events (participants affected / at risk) | 13/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation With Immunosuppression (N=14)
Device related infection (Infections and infestations) | 11 (34)
Pyrexia (General disorders) | 3 (3)
Cytokine release syndrome (Immune system disorders) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hypocalcaemic seizure (Nervous system disorders) | 1 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Systemic immune activation (Immune system disorders) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1)
Cystitis klebsiella (Infections and infestations) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1)
Lower respiratory tract infection fungal (Infections and infestations) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Granuloma skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation With Immunosuppression (N=14)
Hypertension (Vascular disorders) | 10 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6)
Cytokine release syndrome (Immune system disorders) | 5 (6)
Hypothyroidism (Endocrine disorders) | 4 (4)
Urinary tract infection bacterial (Infections and infestations) | 4 (6)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Pyrexia (General disorders) | 4 (5)
Alanine aminotransferase increased (Investigations) | 4 (5)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Sinus bradycardia (Cardiac disorders) | 3 (4)
Occult blood positive (Investigations) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 3 (3)
Ear infection (Infections and infestations) | 2 (2)
Fungal skin infection (Infections and infestations) | 3 (3)
Urinary tract infection enterococcal (Infections and infestations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eye infection bacterial (Infections and infestations) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1)
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Blood bicarbonate decreased (Investigations) | 2 (2)
Blood chloride decreased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2)
Blood urea increased (Investigations) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (2)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (2)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Cystitis klebsiella (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1)
Viral diarrhoea (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Blood immunoglobulin E increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 1 (1)
Red blood cell morphology abnormal (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Disaccharidase deficiency (Metabolism and nutrition disorders) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1)
Nephrocalcinosis (Renal and urinary disorders) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Bilateral breast buds (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphorrhoea (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes